CLINICAL TRIAL: NCT00345657
Title: Extended-Release Niacin/Lovastatin Versus Usual Care for Treatment of Dyslipidemia in a Primary Care Setting (EXTEND Study)
Brief Title: Efficacy Study of Extended-Release Niacin/Lovastatin Versus Usual Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: In His Image (Other)
Collaborators: Kos Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHI-A001
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2006-06-28 (Estimated); Status verified 2006-06

CONDITIONS: Hyperlipidemia; Mixed Hyperlipidemia; Dyslipidemia
Keywords: Hyperlipidemia; Dyslipidemia; Niacin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Combination lipid therapy; Lovastatin
MeSH Terms: conditions — Hyperlipidemias; Hyperlipoproteinemia Type II; Dyslipidemias | interventions — Lovastatin

INTERVENTIONS:
Drug: Niacin Extended Release/Lovastatin

SUMMARY:
The purpose of this study is to investigate the benefits of combination niacin ER/lovastatin in patients receiving standard care who are not at LDL goal per ATP III guidelines.

DETAILED DESCRIPTION:
Both LDL and HDL are important contributors in the pathophysiology of atherosclerosis and coronary artery disease (CAD); however, HDL is often ignored in primary care. The combination of niacin extended-release (ER)/lovastatin in a single tablet formulation (Advicor®) may be the most effective therapeutic option for simultaneously correcting both of these lipoprotein abnormalities to reduce CAD risk. The purpose of this study is to investigate the benefits of combination niacin ER/lovastatin in patients receiving standard care who are not at LDL goal per ATP III guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old with CAD or risk factors for CAD
2. under standard care at Family Medical Care of Tulsa
3. not at LDL goal per ATP III guidelines

Exclusion Criteria:

1. pregnancy/lactating
2. liver disease
3. allergies to statin or niacin
4. active peptic ulcer disease
5. previous treatment with combination therapy for dyslipidemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-07; Study Completion 2004-05

PRIMARY OUTCOMES:
Lipid parameter change at 3 and 6 months
Percent of patients achieving ATP III LDL goals at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Logan, MD, Principal Investigator — In His Image Family Medicine Residency; Edward Rylander, MD, Study Chair — In His Image Family Medicine Residency
Locations (1):
- Family Medical Care of Tulsa, Tulsa, Oklahoma, United States